CLINICAL TRIAL: NCT07362888
Title: A First-in-Human, Phase 1a/1b, Open-Label Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of the Antibody Drug Conjugate ADCE-B05 in Patients With Advanced Solid Tumors
Brief Title: First-in-Human Study of ADCE-B05 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adcendo ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCE-B05-001
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors (Phase 1)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCE-B05 (Experimental): Dose escalation followed by a dose expansion phase. ADCE-B05 is administered intravenously on a 3 weekly dosing cycle
  Interventions: Drug: ADCE-B05

INTERVENTIONS:
Drug: ADCE-B05 — Biological: Antibody-drug conjugate (ADC)

SUMMARY:
The main purpose of the study is to determine the Maximum Tolerated Dose (MTD), the Recommended Expansion Dose and the safety and tolerability of ADCE-B05 when given as a single therapy over a range of different dose levels.

DETAILED DESCRIPTION:
Safety and tolerability will be evaluated by incidence of DLTs. Efficacy will be evaluated by antitumor activity: ORR, DOR, PFR, and TTR per RECIST v 1.1

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of solid tumor
* Advanced disease (i.e., unresectable locally advanced or metastatic) and refractory to, intolerant of, or ineligible for approved therapies
* Radiologically or clinically determined progressive disease during or after most recent line of therapy
* Measurable disease per RECIST 1.1
* ECOG performance status of 0 or 1
* Adequate hematological and biochemical parameters
* A male patient must agree to use barrier contraception during the treatment period and for at least 4 months after the last infusion of study treatment, and refrain from donating sperm during this period. Male patients with a pregnant partner must practice sexual abstinence or use a barrier method of contraception (e.g., condom) to prevent exposure of the fetus or neonate
* A female patient who is not pregnant, not breast feeding, and either not a woman of childbearing potential (WOCBP) or agrees to follow the contraceptive guidance during the treatment period and for at least 7 months after last infusion of study treatment

Exclusion Criteria

* Treatment with systemic anticancer therapy, including any investigational agent within 3 weeks or 5 half-lives (whichever is shorter) prior to study treatment administration
* Prior treatment with an ADC containing a topoisomerase I inhibitor payload
* Primary brain malignancy or known, untreated central nervous system (CNS) or leptomeningeal metastases, or symptoms suggesting CNS involvement for which treatment is required
* Other malignancy
* Major surgical procedure or significant traumatic injury within 28 days prior to study drug administration
* Ongoing systemic infection requiring treatment with antibiotics, antivirals, or antimycotics, other than prophylactic treatment
* Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1
* Clinically significant cardiovascular disease
* Acute infection with human immunodeficiency virus (HIV)-1 or HIV-2
* Current active liver disease due to hepatitis B or hepatitis C
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis or pulmonary lymphangitic carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-03-14 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD/maximum administered dose of ADCE-B05 | From enrollment to the end of Phase 1a (Approximately 11 months after enrollment)
  Incidence of dose-limiting toxicities (DLTs)
Assess the safety and tolerability of ADCE-B05 | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Nature, incidence, severity, and causality of treatment-emergent adverse events (TEAEs) and changes from baseline in laboratory parameters using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0).
  Tolerability as assessed by TEAEs leading to dose interruption, reduction and/or discontinuation

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The maximum concentration (Cmax) will be assessed to characterize the Pharmacokinetic profile of ADCE-B05
Time to maximum concentration (Tmax) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The time to maximum concentration (Tmax) will be assessed to characterize the Pharmacokinetic profile of ADCE-B05
Terminal half-life (T[1/2]) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The terminal half-life (T[1/2]) will be assessed to characterize the Pharmacokinetic profile of ADCE-B05
Area under the concentration-time curve (AUC) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The area under the concentration-time curve (AUC) will be assessed to characterize PK profile of ADCE-B05
Total antibody (TAb) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The total antibody will be assessed to characterize the Pharmacokinetic profile of ADCE-B05
Free (de-conjugated) payload | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  The free (de-conjugated) payload will be assessed to characterize PK profile of ADCE-B05
Objective response rate (ORR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Objective response rate (ORR) will be assessed by Investigator per RECIST v1.1 to evaluate preliminary antitumor activity
Duration of response (DOR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Duration of response DOR will be assessed by Investigator per RECIST v1.1 to evaluate preliminary antitumor activity
Progression-free survival (PFS) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  Progression-free survival (PFS) will be assessed by Investigator per RECIST v1.1 to evaluate preliminary antitumor activity
Disease Control Rate (DCR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  DCR will be assessed by investigator per RECIST v1.1 to evaluate preliminary antitumor activity
Time to Response (TTR) | Throughout the trial duration, completion expected approximately 18 months from completed enrollment
  TTR will be assessed by Investigator per RECIST v1.1 to evaluate preliminary antitumor activity

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Highlands Oncology Group, Springdale, Arkansas
  - Yale University, New Haven, Connecticut
  - University Of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Monash Health, Clayton, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria